CLINICAL TRIAL: NCT06518889
Title: Medium to Long-term Outcomes After Selective Dorsal Rhizotomy in Ambulatory Children and Young People With Cerebral Palsy: A Mixed-methods Study
Brief Title: Medium to Long Term Outcomes of Selective Dorsal Rhizotomy
Acronym: MOSAiC
Status: Recruiting | Type: Observational
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 22BI09
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Cerebral Palsy
Keywords: Selective Dorsal Rhizotomy; Rehabilitation; Physiotherapy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Selective Dorsal Rhizotomy — Selective Dorsal Rhizotomy (SDR) is an irreversible neurosurgical procedure where 50-70% of the sensory nerve roots are cut at the spinal level. The procedure is used to reduce lower limb spasticity permanently and is augmented by intensive rehabilitation for at least two years after surgery to optimise outcomes.

SUMMARY:
The main purpose of this study is to investigate the medium to long-term outcomes (3-10 years) after Selective Dorsal Rhizotomy (SDR) in ambulatory children and young people with cerebral palsy.

The participants will complete a survey, come to hospital for some measurements and tests.

Some parents and children and young people will also be invited to take part in an interview to understand their experiences of SDR.

DETAILED DESCRIPTION:
The aim of this study is to investigate medium (3-5 years) to long-term (6-10 years) outcomes after SDR surgery in ambulatory children with CP and explore how it affects families' (CYP's and parents') lives over time.

A convergent parallel mixed methods study has been designed across two work packages (WPs), which will run in parallel. The International Classification of Functioning, Disability and Health (ICF) will be used as a theoretical framework to guide the data collection and to integrate data from each WP. WP-1 is an observational cohort study and WP-2 is a qualitative study.

In the observational cohort study (WP-1), routinely collected standardised outcome measures will be repeated at one additional time point, more than three years after surgery. This will mirror previous assessments carried out as part of the SDR clinical pathway, which normally concludes two years after surgery. A survey including validated Patient Reported Outcome Measures (PROMs) and a study-specific questionnaire will also be administered in WP-1. The qualitative study (WP-2) will involve an in-depth exploration of parents' and CYPs' views through semi-structured interviews to explore parents' and CYPs' experiences, reflections, and perceptions of outcomes and satisfaction of SDR in relation to previous expectations.

The results from the two WPs will be combined by comparing and contrasting findings from both WPs to provide a more holistic understanding and gain deeper insights into longer-term SDR outcomes. Findings will be used to create evidence-based family resources and decision aids to help families decide whether SDR surgery is the right treatment choice for the child and support their preparation and adjustments after SDR.

ELIGIBILITY:
Inclusion Criteria:

* Children and young people with cerebral palsy (CYPwCP)
* Classified as GMFCS level II and III (ambulatory)
* Aged between 2-15 years at the time of surgery
* Underwent SDR surgery at Great Ormond Street Hospital for Children (GOSH) (between 2013- 2021)
* Had baseline (pre-surgery) assessment and at least one follow-up assessment at 6, 12 or 24 months post-SDR

Parents of CYP with CP who have undergone SDR surgery (and meet the above criteria for CYP)

Exclusion Criteria:

* Children with CP classified as GMFCS level IV, V (non-ambulatory)
* Have any unrelated musculoskeletal problems, such as a recent acute injury

Ages: 7 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children and young people with cerebral palsy who had SDR surgery at Great Ormond Street Hospital (GOSH)
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Function Measure (GMFM) | Single time-point at the follow-up.
  It is a clinical tool designed to evaluate changes in gross motor function in children with cerebral palsy. Performance-based observational tool
Cerebral Palsy Quality of Life (CPQoL) | Single time-point; Parent and CYP questionnaire included in the online survey
  It is a validated tool designed to assess the Quality of Life for children with cerebral palsy across a variety of domains including social wellbeing and acceptance, feelings about functioning, participation and physical health, emotional wellbeing and self-esteem, access to services, pain and impact of disability, and family and parent health.
6- Minute Walk Test | Single time-point at the follow-up.
  Used to test walking capacity and endurance in children with cerebral palsy. Children use their usual walking aids, footwear and orthoses.
Functional Mobility Scale (FMS) | Single time-point; Parent and CYP questionnaire included in the online survey
  The FMS is a performance measure, classifying mobility on the basis of the use of mobility devices across three distances, 5m, 50m, and 500m, which represent home, school, and community distances. The mobility of the child is scored from 1 to 6 for each distance, with 1 representing use of a wheelchair and 6 representing independence on all surfaces.

SECONDARY OUTCOMES:
Modified Ashworth Scale (MAS) | Single time-point at the follow-up.
  This scale is used to measure muscle tone where a leg in moved fast passively in the available range.
Edinburgh Visual Gait Analysis Scale (EVGS) | Single time-point at the follow-up.
  An observational tool to measure gait quality
Gait Outcome Assessment List questionnaire (GOAL) | Single time-point; CYP questionnaire included in the online survey
  The Gait Outcomes Assessment List (GOAL) questionnaire is used to evaluate gait priorities and functional mobility for ambulant children with CP. Scores are additive to provide the item score. Scores for each domain and for the total GOAL are standardized and range from 0 (worst) to 100(best).
  Standardized item, domain, and total GOAL scores are calculated for each child. The maximum total GOAL score is 100 and a higher GOAL score equates to higher function.
Functional Assessment Questionnaire (FAQ) | Single time-point; included in the online survey
  The FAQ is a 10-point scale of the typical level of a child's walking function in their community environment. The walking scale is scored from 1 'cannot take any steps at all' to 10'walks, runs and climbs on level and uneven terrain without difficulty or assistance'. The FAQ is a measure of performance.
Selective Motor Control (SMC) | Single time-point at the follow-up.
  Grading of selective ankle dorsiflexion movement at the ankle ( 0 to 4 scale)
Timed Up and Go (TUG) | Single time-point at the follow-up.
  A functional dynamic balance test. The time taken for the child to stand up from a chair, walk 3 m, turn around, walk back, and sit down is recorded.
The Medical Research Council (MRC) Scale for Testing Muscle Strength | Single time-point at the follow-up.
  0 to 5 grading

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Main, Principal Investigator — Great Ormond Street Institute of Child Health, University College London
Locations (1):
- Great Ormond Street Hospital for Children, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chugh D, Kilbride C, Gimeno H, Aquilina K, Alderson L, Theologis T, Main E. Mixed-methods study exploring medium to longer-term outcomes following selective dorsal rhizotomy in ambulatory children with cerebral palsy at a tertiary hospital in the UK: MOSAiC study protocol. BMJ Open. 2025 Dec 8;15(12):e108558. doi: 10.1136/bmjopen-2025-108558. PMID 41365584